CLINICAL TRIAL: NCT02464514
Title: Investigation of the Developmental, Nutritional and Hormonal Regulation of Ghrelin in Children With Prader-Willi Syndrome (PWS) and Children With Hypothalamic-Derived Obesity: Macronutrient Regulation Sub-study
Brief Title: Macronutrient Regulation of Ghrelin and Peptide YY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Canadian Institutes of Health Research (CIHR) (Other Government); Foundation for Prader-Willi Research (Other); Stollery Children's Hospital Foundation (Other); Alberta Diabetes Institute (Other); Sarah W. Stedman Nutrition and Metabolism Center (Unknown); American Diabetes Association (Other); Duke Children's Miracle Network (Unknown); National Center for Research Resources (NCRR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 5028; 1K23RR021979 (NIH)
Record Dates: First submitted 2015-06-01; First posted 2015-06-08 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2015-06

CONDITIONS: Obesity; Prader Willi Syndrome
Keywords: Obesity; Orexigen; Insulin; Leptin; Adiponectin; Growth hormone replacement
MeSH Terms: conditions — Obesity; Prader-Willi Syndrome; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Healthy obese children (Other): High carbohydrate meal High fat meal
  Interventions: Other: High carbohydrate meal; Other: High fat meal
- Children with Prader Willi Syndrome (Other): High carbohydrate meal High fat meal
  Interventions: Other: High carbohydrate meal; Other: High fat meal

INTERVENTIONS:
Other: High carbohydrate meal — 65% carbohydrate, 17% protein, and 18% fat
Other: High fat meal — 58% fat, 17% protein, and 25% carbohydrate

SUMMARY:
The hyperghrelinemia of children with PWS provides a unique model by which to explore the hormonal and metabolic effects of orexigenic hormones in normal and pathologic conditions. An important question to be addressed by this proposed research includes the macro-nutrient regulation of ghrelin and PYY in obese children and children with PWS. As ghrelin antagonists are considered potential future anti-obesity agents, it is essential to gain understanding of the developmental, nutritional and hormonal regulation of this important orexigenic hormone in children.

DETAILED DESCRIPTION:
Obesity continues to be a prevalent health concern affecting every race of the American population. Studies show that obese children are likely to become obese adults. Also, recent studies report significant years of life lost due to the impact of being an obese adult . Thus, insights into the pathogenesis of childhood obesity and preventative measures are needed to combat the inevitable increase in worldwide incidence of obesity and its associated co-morbidities.

Ghrelin is a 28 amino acid acylated peptide which is an endogenous ligand of the growth hormone secretagogue receptor (GHS-R), a hypothalamic G-protein-coupled receptor. Enteroendocrine cells (X/A-like cells) of the stomach are the major site of ghrelin synthesis, although a minor proportion of ghrelin synthesis occurs in other sites such as the hypothalamus, pituitary, duodenum, jejunum and lung. Secreted in response to meals, ghrelin stimulates feeding through activation of anabolic neurons in the hypothalamic arcuate nucleus that co-express neuropeptide Y (NPY) and agouti-related protein (Agrp). Ghrelin relays its information from the GI tract to specific nuclei in the hypothalamus via the gastric afferent vagal nerve.

Studies in rodents support the premise that ghrelin is involved in energy balance. In humans, physiological levels of ghrelin influence energy homeostasis in humans.The rise in plasma ghrelin concentrations during fasting may play a role in meal initiation and body weight regulation.

Nearly all other forms of obesity are associated with low ghrelin levels. Paradoxically, researchers discovered that ghrelin levels in adults and children with PWS are 3-5 times higher than those in age- and BMI-matched controls. Hyperghrelinemia may thus play a causal role in the hyperphagia and obesity of PWS.

The hyperghrelinemia of children with PWS provides a unique model by which to explore the hormonal and metabolic effects of orexigenic hormones in normal and pathologic condtions. An important question to be addressed by this proposed research includes the macro-nutrient regulation of ghrelin in normal children and children with PWS. As ghrelin antagonists are considered potential future anti-obesity agents, it is essential to gain understanding of the developmental, nutritional and hormonal regulation of this important orexigenic hormone in children.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of PWS confirmed by chromosome analysis (i.e. interstitial deletion of paternally-derived chromosome 15Q, uniparental maternal disomy or other chromosome 15 abnormalities) or normal control
2. Subjects with simple obesity
3. Ages 5 years to 17 years
4. Written informed consent and assent obtained and willingness to comply with the study schedule and procedures.
5. Free T4, TSH values in the normal range (either endogenous or with thyroxine replacement)

Exclusion Criteria:

1. Patients with any other clinically significant disease that would have an impact on body composition including diabetes mellitus, chronic inflammatory bowel disease, chronic severe liver or kidney disease or neurologic disorders
2. Concomitant use of an investigational drug in the past year
3. Patients with an active malignancy
4. Parent or legal guardian unable to provide informed consent.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2004-01; Primary Completion 2005-12 (Actual); Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Change in ghrelin levels | 4 hours
  The change in ghrelin levels will be measured before and after meal consumption in children with PWS, and healthy obese controls. Following an overnight 8 hour fast, subjects will be given either a high carbohydrate or high fat meal. Subjects will be allowed 25 minutes to consume everything on their food tray. Blood samples will be obtained before the meal (fasting) and every 30 minutes thereafter for 4 hours.
Change in PYY concentrations | 4 hours
  The change in PYY concentration levels will be measured before and after meal consumption in children with PWS, and healthy obese controls. Following an overnight 8 hour fast, subjects will be given either a high carbohydrate or high fat meal. Subjects will be allowed 25 minutes to consume everything on their food tray. Blood samples will be obtained before the meal (fasting) and every 30 minutes thereafter for 4 hours.

SECONDARY OUTCOMES:
Fasting Insulin-like growth factor 1 (IGF-1) levels | Baseline
  Baseline Insulin-like growth factor 1 (IGF-1) levels will be measured fasting before the meal in children with PWS, and healthy obese controls
Neuropeptide Y (NPY) | Baseline
  Baseline Neuropeptide Y (NPY) levels will be measured fasting before the meal in children with PWS, and healthy obese controls
Gastric inhibitory polypeptide (GIP) | Baseline
  Baseline Gastric inhibitory polypeptide (GIP) levels will be measured fasting before the meal in children with PWS, and healthy obese controls
Glucagon-like peptide-1 (GLP-1) | Baseline
  Baseline Glucagon-like peptide-1 (GLP-1) levels will be measured fasting before the meal in children with PWS, and healthy obese controls

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Haqq, MD, Principal Investigator — University of Alberta; Michael Freemark, MD, Study Director — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Derived] Gumus Balikcioglu P, Balikcioglu M, Muehlbauer MJ, Purnell JQ, Broadhurst D, Freemark M, Haqq AM. Macronutrient Regulation of Ghrelin and Peptide YY in Pediatric Obesity and Prader-Willi Syndrome. J Clin Endocrinol Metab. 2015 Oct;100(10):3822-31. doi: 10.1210/jc.2015-2503. Epub 2015 Aug 10. PMID 26259133